CLINICAL TRIAL: NCT04164667
Title: Enhancing Executive Function and Self-regulation Success Through the Promotion of Brain Health Behaviors: a Telehealth Pilot Study for Veterans with Chronic Multi-symptom Illness.
Brief Title: Telehealth Pilot for Veterans with Chronic Multi-Symptom Illness.
Acronym: Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: War Related Illness and Injury Study Center (U.S. Federal Agency)
Collaborators: Georgetown University (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01880
Record Dates: First submitted 2019-11-05; First posted 2019-11-15 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Chronic Multisymptom Illness
Keywords: Telehealth; Veterans; Exercise; Meditation; Health Coaching
MeSH Terms: conditions — Motor Activity | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Directed MAP (dMAP) (Experimental): Participants received weekly text message directions from the ANNIE VA messaging system. The directed text messaging system provided details on which app-based meditation and exercise sessions to complete.
  Interventions: Behavioral: Mental and physical (MAP) training intervention
- Self-Guided MAP (sgMAP) (Active Comparator): Participants received the intervention goals at the beginning of the study which included instruction on how to perform each of the individual components of the MAP protocol and how to use the study devices/apps, but they did not receive any further guidance during the intervention.
  Interventions: Behavioral: Mental and physical (MAP) training intervention

INTERVENTIONS:
Behavioral: Mental and physical (MAP) training intervention — In this study, the MAP intervention consisted of two MAP training sessions and one health coaching session per week for eight weeks. Both groups received the same MAP intervention with the exception of the delivery format (directed versus self-guided).
  Each MAP training session included 30 minutes of guided meditation and 30 minutes of moderate-to-vigorous aerobic exercise.
  Other Names: MAP training

SUMMARY:
The objective of this pilot study is to examine the feasibility, safety, and acceptability of a telehealth meditation and physical activity (MAP) intervention among Veterans with chronic multi-symptom illness.

DETAILED DESCRIPTION:
This pilot study innovatively merges with ongoing clinical practice at the War Related Illness and Injury Study Center to explore the utility of new VA technologies and distance-bridging approaches for administering a remote intervention that promotes health behaviors (e.g., physical activity and meditation, called mental and physical training or MAP). Not only does this study intend to examine the feasibility of using these tools within the home setting and integrating these practices into the weekly lives of Veterans, but it also aims to determine the best way to administer this type of intervention by comparing a directed MAP (dMAP) intervention arm to a self-guided MAP (sgMAP) intervention arm. Understanding how much guidance to provide Veterans during their path towards recovery is important since we hope that this pilot study will offer not only evidence that these practices can be administered without supervision but also reveal that giving Veterans the right tools (exercise and meditation app on tablet), guidance (directed text message or holistic goals), and support (video-chat health coaching) can have measurable benefits on symptom severity and function.

ELIGIBILITY:
Inclusion Criteria:

* Previously deployed Veterans
* Experiencing Chronic Multisymptom Illness defined using the Fukuda criteria.
* Able to engage in physical activity
* Has a smart phone
* Co-enrolled in the WRIISC Data Repository Study

Exclusion Criteria:

* Excessive alcohol consumption (AUDIT Score >= 4 (men); AUDIT Score >= 3 (women))
* Current or previous drug use past 90 days.
* Current prominent suicide or homicidal ideation
* Recent exposure to trauma
* Acute or unstable illness
* Dementia or significant cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Feasibility (Recruitment rate) | Through study completion, an average of 6 months
  Recruitment rate was calculated as the number of participants who consented into the study divided by the number of eligible WRIISC patients who were approached during enrollment.
Feasibility (Retention rate) | Through study completion, an average of 6 months
  Retention rate was calculated for each time point (endpoint and 3m follow-up) and reported as a percentage.
Feasibility (Adherence rate) | Through study completion, an average of 6 months
  Due to the multiple components of the intervention, adherence rates were calculated for the meditation and exercise components separately and overall adherence to the MAP training protocol.
Safety of administering a telehealth MAP intervention | Through study completion, an average of 6 months
  Number of adverse events reported during the intervention
Acceptability | Through study completion, an average of 6 months
  Acceptability was quantified using the qualitative feedback provided by participants during their health coaching sessions.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | Baseline to Endpoint (2 months) and baseline to 5 months.
  The BRIEF-A was used to assess executive function across nine overlapping domains: Emotional Control, Initiate, Inhibit, Organization of Materials, Plan/Organize, Self-Monitor, Shift, Task Monitor, and Working Memory. In addition, the Global Executive Composite score and two summary index scores (Behavioral Regulation Index and Metacognition Index) were calculated. Higher scores are indicative of greater difficulty.
Patient Health Questionnaire- Depression scale (PHQ-9) | Baseline to Endpoint (2 months) and baseline to 5 months.
  The PHQ-9 was used to assess the severity of depression symptoms. Higher scores are indicative of greater depression symptoms.
Posttraumatic Symptom Checklist - Military version (PCL-M) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To evaluate the severity of PTSD symptoms in an individual who has had military experience. Higher scores are indicative of greater PTSD symptoms.
Perceived Stress Scale (PSS) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To measure the perception of stress
Brief Symptom Inventory (BSI) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To evaluate the degree of psychological distress.
Five-Factor Mindfulness Questionnaire (FFMQ) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To evaluate mindfulness across five domains: Awareness, Describing, Non-judging of Inner Experience, Non-reactivity to Inner Experience, and Observing.
Medical Outcomes Study Short-Form-36 version 2 (SF-36v2) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To assess quality of life (physical and mental).
Cognitive Difficulties Scale (CDS) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To assess cognitive complaints.
Pittsburgh Sleep Quality Index (PSQI) | Baseline to Endpoint (2 months) and baseline to 5 months.
  To measure the quality and patterns of sleep in adults. Higher scores are indicative of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Reinhard, PsyD, Principal Investigator — DC WRIISC Director; Michelle Costanzo, PhD, Principal Investigator — DC WRIIISC Research Director
Locations (1):
- Washington DC Veteran's Affair Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breneman CB, Pollin K, Chun T, Crock L, Jachimowicz W, McCullers RA, Brewster RC, Alaoui A, Belouali A, Roy MJ, Reinhard MJ, Costanzo ME. Determining the feasibility and acceptability of a randomized telehealth pilot study for veterans with chronic multisymptom illness. Pilot Feasibility Stud. 2025 Apr 9;11(1):43. doi: 10.1186/s40814-025-01628-2. PMID 40205557